CLINICAL TRIAL: NCT04667156
Title: A Single-centre, Single Dose, Randomized, Open-label, Three Period, Six Sequence, Cross Controlled Study to Assess the Relative Bioavailability of the New and Traditional Formulations on SHR6390 in Healthy Subjects
Brief Title: Study to Investigate Relative Bioavailability of Different Formulations of SHR6390 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SHR6390-I-112
Record Dates: First submitted 2020-12-02; First posted 2020-12-14 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Intervention: Drug: SHR6390 new formulation 1(T1) in the first period; SHR6390 new formulation 2 (T2) in the second period; SHR6390 traditional formulation (R) in the last period
  Interventions: Drug: SHR6390
- Sequence 2 (Experimental): Intervention: Drug: SHR6390 traditional formulation (R) in the first period; SHR6390 new formulation 1 (T1) in the second period; SHR6390 new formulation 2 (T2) in the last period
  Interventions: Drug: SHR6390
- Sequence 3 (Experimental): Intervention: Drug: SHR6390 new formulation 2(T2) in the first period; SHR6390 traditional formulation (R) in the second period; SHR6390 new formulation 1 (T1) in the last period
  Interventions: Drug: SHR6390
- Sequence 4 (Experimental): Intervention: Drug: SHR6390 new formulation 1(T1) in the first period; SHR6390 traditional formulation (R) in the second period; SHR6390 new formulation 2 (T2) in the last period
  Interventions: Drug: SHR6390
- Sequence 5 (Experimental): Intervention: Drug: SHR6390 new formulation 2(T2) in the first period; SHR6390 new formulation 1 (T1) in the second period; SHR6390 traditional formulation (R) in the last period
  Interventions: Drug: SHR6390
- Sequence 6 (Experimental): Intervention: Drug: SHR6390 traditional formulation (R) in the first period; SHR6390 new formulation 2 (T2) in the second period; SHR6390 new formulation 1 (T1) in the last period
  Interventions: Drug: SHR6390

INTERVENTIONS:
Drug: SHR6390 — SHR6390 new formulation 1(T1) , SHR6390 new formulation 2 (T2) and SHR6390 traditional formulatin were given in a single dose over three cycles

SUMMARY:
The purpose of this study is to investigate relative bioavailability during the new and traditional formulations of SHR6390 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Execute an informed consent;
2. Male or female aged 18-45 years (including threshold) on the date of signing the informed consent;
3. Male body weight ≥ 50 kg, female body weight ≥ 45 kg, body mass index (BMI) in the range of 19.0-26.0 kg / m2 (including the critical value);
4. Physical examination, vital signs, laboratory examination , 12-Lead ECG, abdominal B-ultrasound, chest X-ray, etc. are normal or abnormal, but the researcher has no clinical significance according to NCI CTCAE 5.0 standard;
5. Fertile subjects had no family planning and had to take acceptable contraceptive measures and no plans to donate eggs and sperm within 7 months from the date of signing informed consent to the last medication; the serum pregnancy test of fertile women within 72 hours before the first administration of the study drug should be negative.

Exclusion Criteria:

1. Those who have previously suffered from primary diseases of important organs, including but not limited to neuropsychiatric, cardiovascular, digestive tract, respiratory system, urinary, endocrine, blood, immune and other diseases, which are judged by the researchers to be unsuitable for the trial;
2. Patients who have received any previous operation affecting gastrointestinal absorption;
3. Patients who had received any surgery within 6 months before screening, or planned to undergo surgery during the study period;
4. Those who lost blood or donated more than 400 ml or received blood transfusion within 3 months before screening;
5. HBsAg positive, HCV antibody positive, HIV antibody positive, syphilis antibody positive;
6. History of drug use or drug abuse, or drug screening positive;
7. Smoking and alcohol addict and unable to stop smoking during the test period; those with positive alcohol screening; those with positive nicotine screening;
8. Allergic constitution, including severe drug allergy or drug allergy history; known allergy to shr6390 tablets or its excipients;
9. Having swallowing resistance or disorder, affecting drug absorption;
10. Participated in other clinical trials and taken the study drug within 3 months before taking the study drug for the first time;
11. Inducers or inhibitors of CYP3A4, CYP2C9 and CYP2C8 were taken within 4 weeks before the first administration of study drug;
12. Taking any prescription drug, over-the-counter drug, traditional Chinese medicine or food supplement within 2 weeks before taking the study drug for the first time;
13. Ingestion of grapefruit containing products, fruit juice, food or beverage containing methylxanthine or alcohol within 72 hours before taking the study drug for the first time; taking strenuous exercise; or having other factors affecting the absorption, distribution, metabolism and excretion of drugs;
14. Lactating women;
15. The researchers considered that the subjects had any other factors that were not suitable for the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Fr | Day1~Day35
  Relative bioavailability of the two new formulations on SHR6390
Cmax | Day1~Day35
  Maximum concentration of SHR6390
AUC0-t | Day1~Day35
  Area under the concentration-time curve from time zero to time t of SHR6390
AUC0-∞ | Day1~Day35
  Area under the concentration-time curve extrapolated to infinity of SHR6390

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided